CLINICAL TRIAL: NCT00928993
Title: An Evaluation of Actigraphy as an Indicator of Sleep and Wake in Children
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Collaborators: Philips Respironics (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB00005369
Record Dates: First submitted 2009-06-25; First posted 2009-06-26 (Estimated); Last update posted 2019-12-27 (Actual); Status verified 2019-12

CONDITIONS: Sleep Monitoring
Keywords: actigraphy; polysomnography; pediatrics; sleep; To validate Actigraphy against polysomnography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Main group: pediatric patients receiving overnight sleep study

SUMMARY:
The purpose of this study is to learn how well an instrument called an Actiwatch-2 can determine whether a child is asleep or awake. The Actiwatch-2 (manufactured by Minimitter/Respironics of Bend, Oregon) is the brand name for an actigraphy monitor; that is, a motion sensor that is typically worn on the wrist and looks like a wrist watch. It measures and records the amount of movement a person makes each minute. After being worn overnight, data are transferred from the Actiwatch to a computer, and a program estimates whether a person is awake or asleep by analyzing the recorded movement data. The enrollment target is 80 participants. Although other actigraphy equipment has been used to monitor sleep in children, the Actiwatch-2 has not been validated in the pediatric population.

ELIGIBILITY:
Inclusion Criteria:

* Children (ages 6 months to 18 years) who are undergoing a medically necessary sleep study [polysomnography (PSG)] in the OHSU Sleep Disorders Laboratory
* ASA classification I and II (children in good health)

Exclusion Criteria:

* ASA classification III, IV (children with a chronic or severe disease).
* Children with developmental delay.
* Children born extremely prematurely (before 32 weeks gestation), as these children and their parents may react differently to experimental procedures
* Children who do not speak English or whose parents do not speak English.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: pediatric patients receiving sleep study as part of their standard medical care
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2009-06 (Actual); Primary Completion 2011-05 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Johnson, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Multnomah Pavilion, OHSU, Portland, Oregon, United States